CLINICAL TRIAL: NCT01863563
Title: Hemostatic Control After Adenotonsillectomy- Open Label QuikClot Study.
Brief Title: Safety Study of Quickclot for Bleeding Control After Adenotonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: version 4 September 2012
Record Dates: First submitted 2013-05-01; First posted 2013-05-29 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea, Obstructive
Keywords: tonsillectomy; adenoidectomy; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Quickclot
Oversight: Data Monitoring Committee: No

ARMS (1):
- QuickClot (Experimental): QuickClot sponge will be applied for one minute each site of tonsillectomy and Adenoidectomy.
  Interventions: Device: QuickClot

INTERVENTIONS:
Device: QuickClot — 1 application of treatment to each tonsil/adenoid removal area

SUMMARY:
Hemostasis will be achieved during Pediatric Tonsillectomy/Adenoidectomy with the use of QuickClot.

DETAILED DESCRIPTION:
The Quickclot dressing contains Kaolin, a natural mineral that promotes the body's clotting process. This dressing will be applied for one minute to the area where the tonsils/adenoids were. The investigators are hoping to develop a standard of practice where Quickclot is a key addition for tonsillectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of adenotonsillar hypertrophy causing obstructive sleep disorders

Exclusion Criteria:

* Patients with signs or symptoms of obstructed breathing
* recurrent pharyngitis
* history of bleeding disorder
* history of prior adenotonsillectomy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Derkay, MD, Principal Investigator — EVMS Department of Otolaryngology
Locations (1):
- Children's Hospital of the Kings Daughters, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Tertiary children's hospital enrolled 100 consectutive children
Groups:
- QuickClot: single dose
Period: Overall Study
Arm/Group | QuickClot
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Quickclot
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.8 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 52
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Total Suction Electrocautery Time Required for Hemostasis Will be Recorded as Seconds
Description: After removal of the adenoids, a tonsil pack wrapped in QuikClot will be placed in the nasopharynx. The investigators will then perform tonsillectomy with the Microdebrider. A QuikClot roll will be placed in the tonsil fossa, and pressure applied via tonsil sponge for one minute. The contralateral tonsil will then be addressed with the same technique. The QuikClot adenoid pack is then removed and residual adenoidal bleeding is addressed with suction electrocautery, followed by placement of a second QuikClot adenoid pack. The tonsil rolls are sequentially removed, followed by control of residual hemostasis with suction electrocautery. A second set of tonsil rolls are placed. After adenoid pack is removed from nasopharynx and bleeding controlled, tonsil rolls are removed, followed by suction electrocautery for any residual hemostasis is performed.
Time Frame: at the time of surgery, 1 hour
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Cauterization Time: single dose
Arm/Group | Cauterization Time
Number analyzed (Participants) | 100
seconds
  total cauterization time | 155.3 (59.7)
  adenoid cauterization time | 60.9 (31.5)
  tonsil cauterization time | 94.5 (41.9)

ADVERSE EVENTS:
Time Frame: 10 days post op
Description: SAE/AE anticipated: episodes of bleeding or dehydration requiring medical intervention
Groups:
- Adverse Events: defined as bleeding or dehydration requiring medical intervention
Arm/Group | Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes